CLINICAL TRIAL: NCT01838902
Title: Primaquine's Gametocytocidal Efficacy in Malaria Asymptomatic Carriers Treated With Dihydroartemisinin-piperaquine in The Gambia
Brief Title: Primaquine's Gametocytocidal Efficacy in Malaria Asymptomatic Carriers
Acronym: PRINOGAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCC 1321
Record Dates: First submitted 2013-04-12; First posted 2013-04-24 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Malaria
Keywords: Malaria; Falciparum; Direct membrane feeding; QT-NASBA; Asexual parasite; Asymptomatic carrier; Gametocytocidal, Gametocyte; Transmission blocking; Sexual stage; Primaquine; Dihydroartemisinin; Piperaquine; Gambia; Africa
MeSH Terms: conditions — Malaria | interventions — Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Eurartesim (control) (Other): All participants will receive a complete course of DHA-PPQ (Eurartesim)
  Interventions: Drug: DHA-PPQ
- Primaquine 0.75mg base/kg (Experimental): Participants will be randomized to receive a complete course of DHA-PPQ plus a single dose of PQ at 0.75mg/kg body weight
  Interventions: Drug: DHA-PPQ; Drug: PQ (0.75)
- Primaquine 0.4mg base /kg (Experimental): Participants will be randomized to receive a complete course of DHA-PPQ plus a single dose of PQ at 0.4mg base/kg Body weight
  Interventions: Drug: DHA-PPQ; Drug: PQ (0.4)
- Primaquine 0.2mg base/kg (Experimental): Participants will be randomized to receive a complete course of DHA-PPQ plus a single dose of PQ at 0.2mg base/kg body weight
  Interventions: Drug: DHA-PPQ; Drug: PQ (0.2)

INTERVENTIONS:
Drug: DHA-PPQ — Participants will receive a 3 day course of DHA-PPQ
  Other Names: Eurartesim
Drug: PQ (0.75) — Participants will receive a single dose of PQ at 0.75mg base/kg body weight
  Other Names: Primaquine
  Arms: Primaquine 0.75mg base/kg
Drug: PQ (0.4) — Participants will receive a single dose of PQ at 0.4mg base/kg body weight
  Other Names: Primaquine
  Arms: Primaquine 0.4mg base /kg
Drug: PQ (0.2) — Participants will receive a single dose of PQ at 0.2mg base/kg body weight
  Other Names: Primaquine
  Arms: Primaquine 0.2mg base/kg

SUMMARY:
In this study, the investigators are interested to know if lower doses of Primaquine together with dihydroartemisinin-piperaquine can produce a similar effect of clearing both sexual and asexual parasites in asymptomatic carriers compared to the recommended dose of primaquine but with a decreased risk of haemolysis.

Children (> 1 year) and adults with normal Glucose-6-phosphate dehydrogenase enzyme levels but with asexual Plasmodium falciparum parasites on the day of screening will be invited to take part in this study.

DETAILED DESCRIPTION:
To date, primaquine (PQ), an 8-aminoquinoline, is the only currently registered product able to clear P. falciparum mature gametocytes. However, its use has been and is still limited by its haematological toxicity (haemolytic anaemia), particularly but not exclusively in individuals with glucose-6-phosphate dehydrogenase deficiency (G6PDd), in whom haemolysis can occur after a single PQ dose. Such an effect is dose-dependent. Considering that the current recommended dose was established several decades ago on a small number of experimentally challenged volunteers, it may be possible to obtain the same effect with a lower dose and hence decrease the risk of haemolysis. The proposed study is a four-arm, open label, randomized, controlled trial. G6PD-normal asymptomatic P. falciparum infected individuals identified through population screening will be randomized to receive either a complete course of dihydroartemisinin-piperaquine (DHA-PPQ) alone (control arm) or a complete course of DHA-PPQ plus a single dose of PQ at 3 differing dose strengths (intervention arms), i.e. 0.75mg/kg, 0.4mg base/kg and 0.2mg base/kg.

The study is planned to enroll 1,200 individuals with an asymptomatic malaria infection during the rainy /transmission season (June - December) from villages around the MRC's field stations at Walikunda and Basse in The Gambia. Asymptomatic parasite carriers identified by qualitative (RDT) and quantitative (parasites counts >20/µl by slide microscopy) methods during population screening exercises at the villages will be invited for a written informed consent and further screening to confirm eligibility, including tests for qualitative G6PD enzyme function (fluorescence spot test) and haemoglobin. If eligible, they will be assigned to one of four study arms using a block randomization scheme in a 1:1:1:1 ratio ensuring a balance in enrollment between the four groups. Enrolled participants will receive ACT treatment on days 0, 1 and 2. On day 2, participants allocated to the PQ arms will receive a dose of primaquine based on determined body weight.

Each participant involvement consists of a maximum of 11 visits over a 42 day period after initiation of treatment. The primary end point is the prevalence of P. falciparum gametocyte carriers at day 7, as determined by QT-NASBA.

ELIGIBILITY:
Inclusion Criteria:

Age ≥1 year

* Weight >10 Kg
* P. falciparum mono-infection, density of at least 20 parasites/μL
* Axillary temperature < 37.5ºC
* Resident in the study area and willingness to reside for the duration of the study
* Written informed consent (plus an assent in children >12years of age)

Exclusion Criteria:

* G6PD Deficiency Haemoglobin <8g/dl

  * Known allergy to any of the study medications
  * Known Pregnancy or breastfeeding
  * Clear/documented history of anti-malarial treatment 2 weeks before contact with study team
  * History of blood transfusion in the previous 3 months
  * Any chronic or acute conditions that might interfere with the study as judged by the research clinician
  * History of sickle cell anaemia

Min Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2013-08; Primary Completion 2015-02 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of P. falciparum gametocyte carriers (QT-NASBA) | Day 7
  Proportion of study participants in each arm with P. falciparum gametocyte carriers as determined by quantitative nucleic acid sequence based amplification assay (QT-NASBA)

SECONDARY OUTCOMES:
Prevalence of P.Falciparum gametocytes carriers | Days 3, 10, 14, 28 and 42
  Prevalence of P. falciparum gametocyte carriers on days 3, 10, 14, 28 and 42, as determined by QT-NASBA
Proportion of individuals infectious to mosquitoes (DMFA) | Day 7
  % of individuals whose day 7 blood samples when fed to mosquitoes by direct membrane feeding assay
Haemoglobin change | Day 0 and days 3, 7, 10, 14, 21, 28, 35 and 42
  Mean (±SD) difference in haemoglobin measured between baseline (day 0) and each follow up visit day by study arm
Prevalence of infection (asexual stages) | Day 3
  Proportion of participants carrying asexual forms of P. Falciparum on day 3
Proportion of participants with recurrent infection (PCR adjusted and unadjusted) | Day 7 to Day 42
  % of participants previously negative for parasites with detectable parasite (by microscopy and PCR) in samples after day 7
Occurrence of adverse events (AEs) and serious adverse events (SAEs) | Day 3 to Day 42
  Occurrence of adverse events (AEs) and serious adverse events (SAEs) during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Umberto D'Alessandro, MD, PhD, Principal Investigator — MRC Unit, Fajara The Gambia
Locations (1):
- Medical Research Council Unit (MRC), The Gambia, Fajara, The Gambia

REFERENCES:
- [Derived] Okebe J, Bousema T, Affara M, Di Tanna GL, Dabira E, Gaye A, Sanya-Isijola F, Badji H, Correa S, Nwakanma D, Van Geertruyden JP, Drakeley C, D'Alessandro U. The Gametocytocidal Efficacy of Different Single Doses of Primaquine with Dihydroartemisinin-piperaquine in Asymptomatic Parasite Carriers in The Gambia: A Randomized Controlled Trial. EBioMedicine. 2016 Nov;13:348-355. doi: 10.1016/j.ebiom.2016.10.032. Epub 2016 Oct 23. PMID 27825738
- [Derived] Okebe J, Bousema T, Affara M, DiTanna G, Eziefula AC, Jawara M, Nwakanma D, Amambua-Ngwa A, Van Geertruyden JP, Drakeley C, D'Alessandro U. The gametocytocidal efficacy of primaquine in malaria asymptomatic carriers treated with dihydroartemisinin-piperaquine in The Gambia (PRINOGAM): study protocol for a randomised controlled trial. Trials. 2015 Mar 1;16:70. doi: 10.1186/s13063-015-0597-1. PMID 25887344